CLINICAL TRIAL: NCT07089563
Title: The Effects of Calisthenics and Life Kinetics Exercises on Reaction Time, Balance, and Swimming Performance in Male Swimmers
Brief Title: Effects of Calisthenics and Life Kinetics on Reaction Time, Balance, and Swimming in Male Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Dr. Ebru CEVİZ, Principal Investigator, Bingol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E-33117789-100-182896
Record Dates: First submitted 2025-06-28; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: No Specific Conditions
Keywords: Male swimmers; Calisthenics exercises; Life kinetics exercises; Reaction; Balance; Swimming performance

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the experimental group receiving calisthenics and life kinetics exercises alongside swimming training or the control group continuing swimming training only.
Masking Description: No parties were masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calisthenics Training Group (Experimental): Participants received Calisthenics Training exercises in addition to their regular swimming training for 8 weeks.
  Interventions: Behavioral: Calisthenics Exercise Program
- Life Kinetik Training Group (Experimental): Participants performed the life kinetics exercise program on specific days per week, in addition to their regular swimming training, for a duration of 8 weeks.
  Interventions: Behavioral: Life Kinetik Exercise Program
- Control Group (No Intervention): Participants continued with their regular swimming training only, without any additional interventions.

INTERVENTIONS:
Behavioral: Calisthenics Exercise Program — The exercises were administered twice a week for eight weeks alongside their regular swimming training, with each session lasting approximately 30 minutes. Calisthenics exercise included crunch, reverse crunch, plank, super plank, superman, sumo squat, and squat jump movements.
  Arms: Calisthenics Training Group
Behavioral: Life Kinetik Exercise Program — The exercise program was conducted twice a week for eight weeks alongside regular swimming training, with each session lasting approximately 30 minutes. It included various exercises designed to improve hand-eye coordination, balance, reaction time, and motor control, such as throwing, catching, and dribbling balls with both the right and left hands. Exercises involved catching the ball mid-air or after a bounce, tossing tennis balls simultaneously with both hands, and throwing balls against a wall with different catching techniques and hand usages to provide varied challenges.
  Arms: Life Kinetik Training Group

SUMMARY:
This study investigates the effects of calisthenics and life kinetics exercises on reaction time, balance, and swimming performance in male swimmers. Participants will be divided into two groups: one group will perform these additional exercises alongside their regular swimming training, while the other group will continue only with swimming. The study aims to find out if adding these exercises can improve swimmers' physical and performance abilities. The study lasts 8 weeks, with measurements taken before and after the program.

DETAILED DESCRIPTION:
his study evaluated the effects of an 8-week calisthenics and life kinetics exercise program on reaction time, balance, and swimming performance in male swimmers. Participants were randomly assigned to either an intervention group, performing the exercises alongside regular swim training, or a control group continuing swim training only. Pre- and post-intervention assessments included standardized reaction time tests, balance evaluations using validated tools, and swimming performance measured through timed swim trials. The study determined whether the addition of these exercises led to significant improvements in the swimmers' physical abilities and performance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male students aged between 18 and 25 years
* Enrolled in the Department of Coaching Education, Faculty of Sports Sciences, Bingöl University
* Specialized in swimming and actively participating in regular swimming training
* No musculoskeletal or neurological conditions in the past six months
* Provided written informed consent and voluntarily agreed to participate

Exclusion Criteria:

* Female students
* Participants who miss more than 2 training sessions during the 8-week intervention
* Current or recent (past 6 months) injury or surgery that limits physical activity
* Use of medication affecting balance, coordination, or motor function
* Participation in any other training program outside of the study during the intervention period

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only self-identified males are eligible to participate in the study.
Enrollment: 30 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
15-Meter Freestyle Swimming Time | At baseline and 8 weeks of training
  Participants' performance was assessed using a Selex stopwatch to measure the time (in seconds) taken to swim 15 meters freestyle. Timing started when the swimmer's toes left the starting block and stopped when their head crossed the 15-meter marker. Standard warm-up procedures and competitive swimming rules were followed.
25-Meter Freestyle Swimming Time | At baseline and 8 weeks of training
  The time (in seconds) required to complete a 25-meter freestyle swim was measured using a Selex SLX 508 digital sports stopwatch. Standard warm-up was completed before testing. Participants were instructed to swim at maximal effort.

SECONDARY OUTCOMES:
Reaction Time | At baseline and 8 weeks of training
  Reaction Time (Digital Reaction Test Device) Time Frame: At baseline and after 8 weeks of training Description: Reaction time was measured using a digital reaction test device. In each trial, participants responded to a color change on the screen by touching it as quickly as possible. The test was repeated three times, and the best (shortest) reaction time was recorded in milliseconds (ms).

OTHER OUTCOMES:
Static Balance Score | At baseline and 8 weeks of training
  Static balance was assessed using the Pagani TM stabilometric platform (Elettronica Pagani, Italy). Participants stood barefoot on a 50×50 cm platform surface for 30 seconds in a standardized foot position (30° angle, 2 cm between heels), while focusing on a fixed target at eye level. No external distractions were present during the test.
  The following parameters were recorded through the platform's software:
  * R-LSD (Right-Left Standard Deviation)
  * A-PSD (Anterior-Posterior Standard Deviation)
  * M-LMSV (Medial-Lateral Mean Sway Velocity)
  * A-PMSV (Anterior-Posterior Mean Sway Velocity)
  * CPPL (Center of Pressure Path Length)
  * SA (Sway Area) Each participant performed the test once, and the raw values were used for analysis. All data were collected using a computerized system integrated with the stabilometric platform.
Right-Left Standard Deviation (R-LSD) | At baseline and 8 weeks of training
  Right-left sway was recorded using the Pagani TM stabilometric platform. Higher values indicate poorer balance.
  Unit of Measure: millimeters (mm)
Anterior-Posterior Standard Deviation (A-PSD) | At baseline and 8 weeks of training
  Anterior-posterior sway was recorded using the Pagani TM stabilometric platform. Higher values indicate poorer balance.
  Unit of Measure: millimeters (mm)
Medial-Lateral Mean Sway Velocity (M-LMSV) | At baseline and 8 weeks of training
  The average speed of center of pressure movement in the medial-lateral direction during the balance test. Elevated values indicate greater postural instability.
  Unit of Measure: millimeters per second (mm/s)
Anterior-Posterior Mean Sway Velocity (A-PMSV) | At baseline and 8 weeks of training
  The average velocity of sway in the anterior-posterior direction, calculated from center of pressure data. Higher values represent impaired static balance.
  Unit of Measure: millimeters per second (mm/s)
Center of Pressure Path Length (CPPL) | At baseline and 8 weeks of training
  Total length of the trajectory followed by the center of pressure during the 30-second static balance test. Longer path length indicates greater postural sway and poorer balance control.
  Unit of Measure: millimeters (mm)
Sway Area (SA) | At baseline and 8 weeks of training
  The area covered by the center of pressure trajectory during the test, representing the spatial extent of postural sway. Larger areas suggest reduced postural stability.
  Unit of Measure: square millimeters (mm²)
Dynamic Balance Score | At baseline and 8 weeks of training
  Dynamic balance was assessed using the Libra (EasyTech) balance platform, which includes interchangeable blocks with three difficulty levels: 12 cm (easy), 24 cm (medium), and 40 cm (hard). For this study, the medium difficulty level with the 24 cm block was selected. Participants performed two separate 30-second trials in a double-leg stance, focusing their gaze on a fixed point located 3 meters away. The best result of the two trials was recorded for analysis.
  Seven fundamental balance parameters based on sway area (measured in square millimeters, mm²) and reaction times (measured in milliseconds, ms) were analyzed:
  * DBP (Dynamic Balance Performance)
  * RSA (Right Sway Area)
  * LSA (Left Sway Area)
  * ROSA (Right Outer Sway Area)
  * LOSA (Left Outer Sway Area)
  * RSRT (Right Sway Reaction Time)
  * LSRT (Left Sway Reaction Time)
Dynamic Balance Performance (DBP) | At baseline and 8 weeks of training
  The duration participants were able to maintain balance during the dynamic test on the Libra platform. Shorter durations indicate better balance performance.
  Unit of Measure: seconds (s)
Right Sway Area (RSA) | At baseline and 8 weeks of training
  The area covered by postural sway on the right side during dynamic balance testing. Higher values represent greater instability.
  Unit of Measure: square millimeters (mm²)
Left Sway Area (LSA) | At baseline and 8 weeks of training
  The area covered by postural sway on the left side during dynamic balance testing. Larger sway areas indicate poorer balance performance.
  Unit of Measure: square millimeters (mm²)
Right Outer Sway Area (ROSA) | At baseline and 8 weeks of training
  The extent of sway beyond the central area on the right side. Increased values signify a loss of postural control.
  Unit of Measure: square millimeters (mm²)
Left Outer Sway Area (LOSA) | At baseline and 8 weeks of training
  The extent of sway beyond the central area on the left side during dynamic testing. Higher values reflect reduced balance stability.
  Unit of Measure: square millimeters (mm²)
Right Sway Reaction Time (RSRT) | At baseline and 8 weeks of training
  The time it took for participants to react and stabilize following a perturbation or sway toward the right. Longer times indicate delayed neuromuscular response and impaired dynamic balance.
  Unit of Measure: milliseconds (ms)
Left Sway Reaction Time (LSRT) | At baseline and 8 weeks of training
  The time it took for participants to respond to sway in the left direction during the dynamic balance test. Longer reaction times represent poorer dynamic balance control.
  Unit of Measure: milliseconds (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Harun GENÇ, AssocProfDr, Principal Investigator — Bingöl University Faculty of Sports Sciences
Locations (1):
- Bingöl University, Bingöl, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical considerations and lack of participant consent for public data sharing.